CLINICAL TRIAL: NCT02035501
Title: Treatment of TNNT1-Myopathy With L-Tyrosine. A Double-blind, Placebo-controlled Crossover Trial.
Brief Title: Treatment of TNNT1-Myopathy With L-Tyrosine.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Shimon Edverson, MD, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SimonEdvardson1
Record Dates: First submitted 2013-07-02; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Nemaline Myopathy
MeSH Terms: conditions — Myopathies, Nemaline | interventions — Tyrosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- L-Tyrosine (Active Comparator)
  Interventions: Drug: L-Tyrosine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-Tyrosine
  Arms: L-Tyrosine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate if treatment with L-Tyrosine improves selected outcome measures of TNNT1 myopathy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* any age with TNNT1-related myopathy

Exclusion Criteria:

* Patients who are non-cooperative or parents/ legal guardians who are unwilling to sign consent form

Max Age: 20 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
1. goal attainment score | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel